CLINICAL TRIAL: NCT02549209
Title: Phase II Study of Pembrolizumab in Combination With Carboplatin and Paclitaxel for Advanced or Recurrent Endometrial Adenocarcinoma
Brief Title: Pembro/Carbo/Taxol in Endometrial Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Daniela Matei, MD (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry); Hoosier Cancer Research Network (Other)
Responsible Party: Sponsor-Investigator, Daniela Matei, MD, Sponsor-Investigator, Big Ten Cancer Research Consortium
Organization: Big Ten Cancer Research Consortium (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BTCRC GYN15-013
Record Dates: First submitted 2015-09-11; First posted 2015-09-15 (Estimated); Results first posted 2021-11-30 (Actual); Last update posted 2022-03-02 (Actual); Status verified 2022-02

CONDITIONS: Endometrial Cancer; Endometrial Adenocarcinoma
Keywords: Pembrolizumab; Keytruda; Anti-Programmed [Cell] Death Protein 1 (PD-1) Antibody; Carboplatin; Paclitaxel
MeSH Terms: conditions — Endometrial Neoplasms; Parkinson Disease 4, Autosomal Dominant Lewy Body | interventions — pembrolizumab; Paclitaxel; Carboplatin

STUDY DESIGN:
Masking Description: Open-Label
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Investigational Treatment (Experimental): Subjects with no prior therapy:
  * Pembrolizumab administered at 200 mg
  * Paclitaxel administered at 175mg/m2
  * Carboplatin administered at an AUC of 6
  Subjects with prior external beam radiation therapy (XRT) and/or platinum-based chemotherapy must initiate paclitaxel and carboplatin at a reduced dose:
  * Pembrolizumab administered at 200 mg
  * Paclitaxel administered at 135mg/m2
  * Carboplatin administered at an AUC of 5
  Interventions: Drug: Pembrolizumab; Drug: Paclitaxel; Drug: Carboplatin

INTERVENTIONS:
Drug: Pembrolizumab — Pembrolizumab 200 mg will be administered every 3 weeks for all subjects
  Other Names: MK-3475; Keytruda®
Drug: Paclitaxel — For subjects with no prior therapy, paclitaxel will be dosed at 175mg/m2 and be administered as a 3-hour continuous IV infusion.
  Subjects with prior XRT/platinum-based chemotherapy must initiate paclitaxel at 135mg/m2 and be administered as a 3-hour continuous IV infusion.
  Other Names: Taxol®
Drug: Carboplatin — For subjects with no prior therapy, carboplatin will be dosed at an AUC of 6 and given as an IV infusion in 250ml of D5W over 30 minutes.
  Subjects with prior XRT/platinum-based chemotherapy must initiate carboplatin at an AUC of 5 given as an IV infusion in 250ml of D5W over 30 minutes.
  Other Names: Paraplatin®

SUMMARY:
This is a single-arm, open-label, multi-center phase II study for subjects with measurable advanced or recurrent endometrial cancer using pembrolizumab in combination with carboplatin and paclitaxel chemotherapy. As this combination of agents has not been tested in this subject population, the first six subjects enrolled will constitute a safety run-in cohort.

DETAILED DESCRIPTION:
OUTLINE: This is a multi-center study.

INVESTIGATIONAL TREATMENT:

To ensure the safety of this combination treatment, an initial safety run-in will be conducted for the first 6 subjects. This initial cohort of 6 subjects will be enrolled and treated with standard doses as described below. Based on toxicity analysis of the initial 6 subjects following completion of 18 weeks of treatment, it will be determined if an extended safety run-in period would be beneficial.

In the absence of receiving any prior therapy, eligible subjects will be treated as follows on D1 of cycles lasting 21 days (3 weeks) for a maximum of 6 cycles:

* Pembrolizumab 200mg will be administered as a 30-minute intravenous (IV) infusion every 3 weeks.
* Paclitaxel will be dosed at 175mg/m2 and be administered as a 3-hour continuous IV infusion.
* Carboplatin will be dosed at area under the curve (AUC) of 6 and given as an IV infusion in 250ml of D5W over 30 minutes.

Subjects who have had prior radiotherapy/platinum-based chemotherapy must initiate paclitaxel and carboplatin at the following reduced dose levels if they have had prior external radiotherapy involving the whole pelvis or abdomen or over 50% of their spine, and/or prior platinum-based chemotherapy for this, or any other cancer. Eligible subjects will be treated as follows on Day 1 (D1) of cycles lasting 21 days (3 weeks) for a maximum of 6 cycles:

* Pembrolizumab 200mg administered as a 30-minute intravenous (IV) infusion every 3 weeks.
* Paclitaxel will be dosed at 135mg/m2 and be administered as a 3-hour continuous IV infusion.
* Carboplatin will be dosed at an AUC of 5 and given as an IV infusion in 250ml of D5W over 30 minutes.

Subsequent doses of paclitaxel and carboplatin may be escalated to the higher doses as indicated above, provided these subjects do not exhibit hematologic or nonhematologic toxicity > Grade 1, except alopecia.

The following laboratory values must be obtained within 14 days prior to registration for protocol therapy:

Hematopoietic:

* Hemoglobin (Hgb) > 9 g/dL (without transfusion or erythropoietin (EPO) dependency within 7 days of assessment)
* Platelets > 100 K/mm3
* Absolute neutrophil count (ANC) ≥ 1.5 K/mm3

Renal:

* Creatinine or measured/calculated creatinine clearance (as calculated by institutional standard) ≤ 1.5 X institutional upper limits of normal (ULN) OR ≥60mL/min for subjects with creatinine levels > 1.5 x institutional ULN

Hepatic:

* Serum total bilirubin ≤ 1.5 x upper limit of normal (ULN) OR direct bilirubin ≤ ULN for subjects with total bilirubin levels > 1.5 ULN
* Aspartate aminotransferase (AST), alanine transaminase (ALT) or alkaline phosphatase (ALP) < 2.5 x ULN OR ≤ 5 x ULN for subjects with liver metastases
* Albumin ≥ 2.5 mg/dL

Coagulation (Blood Clotting) Tests:

* International normalized ratio (INR) or prothrombin time (PT) ≤ 1.5 x ULN unless subject is receiving anti-coagulant therapy as long as partial thromboplastin time (PTT) is within therapeutic range of intended use of anticoagulants
* Activated partial thromboplastin time (aPTT) ≤ 1.5 x ULN unless subject is receiving anti-coagulant therapy as long as PT or PTT is within therapeutic range of intended use of anticoagulants

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent and HIPAA authorization for release of personal health information prior to registration for protocol therapy.

  o NOTE: HIPAA authorization may be included in the informed consent or obtained separately.
* Age ≥ 18 years at the time of consent.
* ECOG Performance Status of 0 or 1 within 28 days prior to registration for protocol therapy.
* Histological evidence of newly diagnosed Stage III or IV or recurrent endometrial carcinoma who have had definitive surgery for endometrial cancer (at least hysterectomy and bilateral salpingo-oophorectomy). Pathologic documentation of the recurrence (i.e., biopsy) will be performed per standard of care, at the treating physician's discretion. If a subject with recurrence is undergoing a biopsy for clinical indications and is willing and able, an optional collection of 3 frozen tissue cores of the recurrence site is requested for correlative analysis.
* Measurable disease according to RECIST v1.1 and obtained by imaging within 28 days prior to registration for protocol therapy. Disease in an irradiated field as the only site of measurable disease is acceptable only if there has been clear progression since completion of radiation treatment.
* The subject must have recovered (≤ grade 1) from the acute toxic effects of prior therapy.
* Prior treatment: Subjects may have received none or one platinum-based chemotherapy regimen and none or one non-platinum regimen. Subjects having received prior platinum-based chemotherapy must have a disease-free interval > 6 months (be platinum sensitive).
* Prior therapy with hormones or biologic agents is allowed. These treatments must be discontinued at least 28 days prior to registration for protocol therapy.
* The subject must have completed radiation therapy at least 28 days prior to registration for protocol therapy, provided that toxicity has resolved to ≤ grade 1.

  * NOTES: Subjects may have received prior radiation therapy for treatment of endometrial carcinoma. Prior radiation therapy may have included pelvic radiation therapy, extended field pelvic/para-aortic radiation therapy, and/or intravaginal brachytherapy. Chemotherapy used for radiation sensitization is allowed. Chemotherapy used for radiation sensitization will not count as second chemotherapy regimen.
  * Palliative radiation given primarily for symptom relief, without the intent to treat or cure the patient's endometrial cancer is excluded from the above criteria. Treatment-directed radiation will be defined as more than 30 Gy of radiation.
* No prior malignancy is allowed except for adequately treated basal cell or squamous cell skin cancer, in situ cervical cancer, or other cancer for which the subject has been disease-free for at least 5 years.
* Female subjects must be of non-childbearing potential. Women of childbearing potential are those who have not been surgically sterilized or have not been free from menses for ≥1 year.
* Laboratory values must be obtained within 14 days prior to registration for protocol therapy. Note: Institutional/laboratory upper limit of normal (ULN)
* Hemoglobin (Hgb) > 9 g/dL (without transfusion or EPO dependency within 7 days of assessment)
* Platelets > 100 K/mm3
* Absolute neutrophil count (ANC) ≥ 1.5 K/mm3
* Creatinine or measured/calculated creatinine clearance (as calculated by institutional standard) ≤ 1.5 X institutional ULN OR ≥60mL/min for subjects with creatinine levels > 1.5 x institutional ULN
* Serum total bilirubin ≤ 1.5 ULN OR Direct bilirubin ≤ ULN for subjects with total bilirubin levels > 1.5 ULN
* AST, ALT or alkaline phosphatase < 2.5 ULN OR ≤ 5 x ULN for subjects with liver metastases
* Albumin ≥ 2.5 mg/dL
* International normalized ratio (INR) or prothrombin time (PT) ≤ 1.5 x ULN unless subject is receiving anti-coagulant therapy as long as PTT is within therapeutic range of intended use of anticoagulants
* Activated Partial Thromboplastin Time (aPTT) ≤ 1.5 x ULN unless subject is receiving anti-coagulant therapy as long as PT or PTT is within therapeutic range of intended use of anticoagulants

Exclusion Criteria:

* Subjects with carcinosarcoma.
* Subjects who have a solitary central pelvic recurrence, which can be curatively resected.
* Hypersensitivity to pembrolizumab or any of its excipients.
* Has had a prior anti-cancer monoclonal antibody (mAb) within 4 weeks prior to registration for protocol therapy or who has not recovered (i.e., ≤ Grade 1 or at baseline) from adverse events due to agents administered more than 4 weeks earlier.
* Has known active central nervous system (CNS) metastases and/or carcinomatous meningitis. Subjects with previously treated brain metastases may participate provided they are stable (without evidence of progression by imaging for at least four weeks prior to registration for protocol therapy and any neurologic symptoms have returned to baseline), have no evidence of new or enlarging brain metastases, and are not using steroids for at least 7 days prior registration for protocol therapy. This exception does not include carcinomatous meningitis, which is excluded regardless of clinical stability.
* NOTE: Subjects with neurological symptoms must undergo a head CT scan or brain MRI to exclude brain metastasis.
* Treatment with any investigational agent within 28 days prior to registration for protocol therapy.
* Has known history of Human Immunodeficiency Virus (HIV) (HIV 1/2 antibodies).
* Active autoimmune disease that has required systemic treatment in past 2 years (i.e., with use of disease modifying agents, corticosteroids, or immunosuppressive drugs). Replacement therapy (e.g., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment.
* Has received systemic steroid therapy or any other form of immunosuppressive therapy within 7 days prior to registration for protocol therapy. (Prednisone (or equivalent) < 10mg/ day is allowed).
* Has a known history of active TB (Bacillus Tuberculosis).
* Pulmonary conditions such as sarcoidosis, silicosis, idiopathic pulmonary fibrosis, or hypersensitivity pneumonitis.
* Has a history of (non-infectious) pneumonitis that required steroids or has current pneumonitis.
* Evidence of interstitial lung disease.
* Has an active infection requiring systemic therapy with the exception of an uncomplicated urinary tract infection.
* Pre-existing peripheral neuropathy that is ≥ Grade 2 by CTCAE v4 criteria.
* Has received prior therapy with an anti-PD-1, anti-PD-L1, or anti-PD-L2 agent.
* Has a known history of Hepatitis B (defined as Hepatitis B surface antigen [HBsAg] reactive) or known active Hepatitis C virus (defined as HCV RNA [qualitative] is detected) infection. Note: no testing for Hepatitis B and Hepatitis C is required unless mandated by local health authority.
* Has received a live vaccine within 30 days prior to registration for protocol therapy.

  o NOTE: Seasonal influenza vaccines for injection are generally inactivated flu vaccines and are allowed; however, intranasal influenza vaccines (e.g., Flu-Mist) are live attenuated vaccines, and are not allowed.
* History of solid organ or stem cell transplant requiring immunosuppressive medications.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2017-08-22 (Actual); Primary Completion 2019-12-12 (Actual); Study Completion 2022-02-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Daniela Matei, M.D., Study Chair — Big Ten Cancer Research Consortium
Locations (6):
- United States (6):
  - Ironwood Cancer and Research Centers, Mesa, Arizona
  - Northwestern University, Robert H. Lurie Cancer Center, Chicago, Illinois
  - Northwestern Medicine Lake Forest Hospital, Lake Forest, Illinois
  - Indiana University Melvin and Bren Simon Cancer Center, Indianapolis, Indiana
  - University of Iowa Hospitals and Clinics, Iowa City, Iowa
  - University of Minnesota, Minneapolis, Minnesota

REFERENCES:
- See also: Big Ten Cancer Research Consortium Website — http://www.bigtencrc.org

RESULTS

PARTICIPANT FLOW:
Groups:
- Investigational Treatment: Subjects with no prior therapy:
  * Pembrolizumab administered at 200 mg
  * Paclitaxel administered at 175mg/m2
  * Carboplatin administered at an AUC of 6
  Subjects with prior external beam radiation therapy (XRT) and/or platinum-based chemotherapy must initiate paclitaxel and carboplatin at a reduced dose:
  * Pembrolizumab administered at 200 mg
  * Paclitaxel administered at 135mg/m2
  * Carboplatin administered at an AUC of 5
  Pembrolizumab: Pembrolizumab 200 mg will be administered every 3 weeks for all subjects
  Paclitaxel: For subjects with no prior therapy, paclitaxel will be dosed at 175mg/m2 and be administered as a 3-hour continuous IV infusion.
  Subjects with prior XRT/platinum-based chemotherapy must initiate paclitaxel at 135mg/m2 and be administered as a 3-hour continuous IV infusion.
  Carboplatin: For subjects with no prior therapy, carboplatin will be dosed at an AUC of 6 and given as an IV infusion in 250ml of D5W over 30 minutes.
  Subjects with prior XRT/platinum-based chemotherapy must initiate carboplatin at an AUC of 5 given as an IV infusion in 250ml of D5W over 30 minutes.
Period: Overall Study
Arm/Group | Investigational Treatment
Started | 46
Completed | 46
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Investigational Treatment
Number analyzed (Participants) | 46
Age, Continuous [Median (Full Range); unit: years] | 66 [43 to 86]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 46
  Male | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 3
  White | 39
  More than one race | 0
  Unknown or Not Reported | 3
Region of Enrollment [Number; unit: participants]
  United States | 46
Stage at Diagnosis [Count of Participants; unit: Participants] — International Federation of Gynecology and Obstetrics (FIGO) stage ranges from I through IV where Stage I = cancer is growing inside the uterus. It may also be growing into the glands of the cervix, but not into the supporting connective tissue of the cervix (T1). It has not spread to nearby lymph nodes (N0) or to distant sites (M0) and Stage IVB = cancer has spread to inguinal (groin) lymph nodes, the upper abdomen, the omentum, or to organs away from the uterus, such as the lungs, liver, or bones (M1). The cancer can be any size and it might or might not have spread to other lymph nodes.
  Participants
    IA | 13
    IB | 7
    II | 8
    IIIA | 4
    IIIC1 | 3
    IIIC2 | 3
    IVA | 2
    IVB | 6
Diagnosis Type [Count of Participants; unit: Participants]
  Primary | 12
  Recurrent | 34
Tumor Grade [Count of Participants; unit: Participants] — Tumors are graded as 1, 2, 3, or 4, depending on the amount of abnormality. In Grade 1 tumors, the tumor cells and the organization of the tumor tissue appear close to normal, but Grade 3 and Grade 4 tumors do not look like normal cells and tissue. Grade 3 and Grade 4 tumors tend to grow rapidly and spread faster than tumors with a lower grade.
  Participants
    1 | 14
    2 | 10
    3 | 22
Histology [Count of Participants; unit: Participants]
  Clear Cell | 3
  Endometrioid | 27
  Mucinous | 0
  Other | 5
  Serous | 11
Previous Treatment [Number; unit: participants]
  Carboplatin/paclitaxel | 19
  External beam radiotherapy | 23
  Brachytherapy | 14

OUTCOME MEASURES:

1. Primary Outcome: Objective Response Rates (ORR)
Description: Objective response rate(ORR) is defined as the percentage of subjects with a partial response or complete response according to immune-related RECIST criteria.
  Immune-Related Response Criteria:
  Complete Response(irCR): Disappearance of all lesions in two consecutive observations not less than 4 wk apart.
  Partial Reponse (irPR): decrease in tumor burden ≥50 %relative to baseline confirmed by a consecutive assessment at least 4 wk after first documentation Stable Disease (irSD): not meeting criteria for irCR or irPR, in absence of irPD
Time Frame: From start of treatment Day 1 (D1) and assessed for a maximum of 18 months
Population: Forty-three of the enrolled patients were evaluable for efficacy using the primary endpoint of ORR. Three patients received a single dose of therapy and were not evaluable for response due to transition to hospice care, a severe allergic reaction to therapy, or no further follow up.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Investigational Treatment
Number analyzed (Participants) | 43
percentage of participants | 74.4 [58.8 to 86.5]

2. Secondary Outcome: Proportion of Subjects Who Experience ≥ Grade 3 Toxicity According Per Common Toxicity Criteria for Adverse Effects (CTCAE) v4 Criteria
Description: Proportion of subjects who experience ≥ Grade 3 toxicity regardless of relation according per Common Toxicity Criteria for Adverse Effects (CTCAE) v4 criteria while receiving pembrolizumab in combination with standard carboplatin/paclitaxel therapy
Time Frame: From time of consent to up to a maximum of 7 months(30 days following cessation of treatment )
Measure: Number; unit: proportion of participants
Arm/Group | Investigational Treatment
Number analyzed (Participants) | 46
proportion of participants | 0.74

ADVERSE EVENTS:
Time Frame: From time of consent to up to a maximum of 7 months(30 days following cessation of treatment )
Description: CTCAE grades the severity of an adverse event from 1-5 where 1=least severe and 5=death.
Arm/Group | Investigational Treatment
All-Cause Mortality (participants affected / at risk) | 11/46
Serious Adverse Events (participants affected / at risk) | 16/46
Other Adverse Events (participants affected / at risk) | 46/46
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Investigational Treatment (N=46)
ACUTE KIDNEY INJURY (Renal and urinary disorders) | 1 (1)
ANAPHYLAXIS (Immune system disorders) | 1 (3)
ANEMIA (Blood and lymphatic system disorders) | 1 (1)
ATAXIA (Nervous system disorders) | 1 (1)
COLITIS (Gastrointestinal disorders) | 1 (1)
DEHYDRATION (Metabolism and nutrition disorders) | 2 (2)
DYSPNEA (Respiratory, thoracic and mediastinal disorders) | 1 (2)
FATIGUE (General disorders) | 1 (1)
FEVER (General disorders) | 3 (3)
HEMATOMA (Vascular disorders) | 1 (1)
HYPERTHYROIDISM (Endocrine disorders) | 1 (1)
HYPOKALEMIA (Metabolism and nutrition disorders) | 2 (2)
INFECTIONS AND INFESTATIONS (Infections and infestations) | 1 (1)
MUSCLE WEAKNESS LOWER LIMB (Musculoskeletal and connective tissue disorders) | 1 (1)
NAUSEA (Gastrointestinal disorders) | 1 (1)
NEUTROPHIL COUNT DECREASED (Investigations) | 1 (1)
SYNCOPE (Nervous system disorders) | 2 (2)
THROMBOEMBOLIC EVENT (Vascular disorders) | 1 (1)
UPPER RESPIRATORY INFECTION (Infections and infestations) | 1 (1)
VESTIBULAR DISORDER (Ear and labyrinth disorders) | 1 (1)
VOMITING (Gastrointestinal disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Investigational Treatment (N=46)
ABDOMINAL DISTENSION (Gastrointestinal disorders) | 1 (2)
ABDOMINAL PAIN (Gastrointestinal disorders) | 15 (15)
ACTIVATED PARTIAL THROMBOPLASTIN TIME PROLONGED (Investigations) | 9 (13)
ACUTE KIDNEY INJURY (Renal and urinary disorders) | 2 (2)
AGITATION (Psychiatric disorders) | 3 (4)
ALANINE AMINOTRANSFERASE INCREASED (Investigations) | 7 (8)
ALKALINE PHOSPHATASE INCREASED (Investigations) | 8 (12)
ALLERGIC RHINITIS (Respiratory, thoracic and mediastinal disorders) | 3 (3)
ALOPECIA (Skin and subcutaneous tissue disorders) | 21 (26)
ANEMIA (Blood and lymphatic system disorders) | 36 (92)
ANOREXIA (Metabolism and nutrition disorders) | 12 (19)
ANXIETY (Psychiatric disorders) | 10 (11)
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 11 (14)
ARTHRITIS (Musculoskeletal and connective tissue disorders) | 5 (5)
ASCITES (Gastrointestinal disorders) | 1 (2)
ASPARTATE AMINOTRANSFERASE INCREASED (Investigations) | 10 (11)
BACK PAIN (Musculoskeletal and connective tissue disorders) | 11 (11)
BLADDER SPASM (Renal and urinary disorders) | 1 (1)
BLOATING (Gastrointestinal disorders) | 2 (2)
BLOOD AND LYMPHATIC SYSTEM DISORDERS (Blood and lymphatic system disorders) | 5 (6)
BLOOD BILIRUBIN INCREASED (Investigations) | 3 (5)
BLURRED VISION (Eye disorders) | 4 (4)
BONE PAIN (Musculoskeletal and connective tissue disorders) | 1 (1)
BRONCHIAL INFECTION (Infections and infestations) | 1 (1)
BRUISING (Injury, poisoning and procedural complications) | 5 (6)
CARDIAC DISORDERS (Cardiac disorders) | 1 (1)
CATARACT (Eye disorders) | 1 (1)
CHEST WALL PAIN (Musculoskeletal and connective tissue disorders) | 1 (1)
CHILLS (General disorders) | 3 (4)
CHOLESTEROL HIGH (Investigations) | 5 (5)
CHRONIC KIDNEY DISEASE (Renal and urinary disorders) | 1 (1)
COLITIS (Gastrointestinal disorders) | 1 (1)
COLONIC FISTULA (Gastrointestinal disorders) | 1 (1)
CONFUSION (Psychiatric disorders) | 1 (1)
CONGENITAL, FAMILIAL AND GENETIC DISORDERS (Congenital, familial and genetic disorders) | 1 (1)
CONSTIPATION (Gastrointestinal disorders) | 17 (28)
COUGH (Respiratory, thoracic and mediastinal disorders) | 19 (21)
CREATININE INCREASED (Investigations) | 5 (6)
CYSTITIS NONINFECTIVE (Renal and urinary disorders) | 1 (1)
DEHYDRATION (Metabolism and nutrition disorders) | 4 (6)
DEPRESSION (Psychiatric disorders) | 7 (8)
DIARRHEA (Gastrointestinal disorders) | 22 (32)
DIZZINESS (Nervous system disorders) | 8 (12)
DRY MOUTH (Gastrointestinal disorders) | 1 (1)
DRY SKIN (Skin and subcutaneous tissue disorders) | 4 (4)
DYSGEUSIA (Nervous system disorders) | 6 (8)
DYSPEPSIA (Gastrointestinal disorders) | 2 (2)
DYSPNEA (Respiratory, thoracic and mediastinal disorders) | 17 (25)
EAR PAIN (Ear and labyrinth disorders) | 1 (1)
EDEMA LIMBS (General disorders) | 15 (17)
EDEMA TRUNK (General disorders) | 2 (2)
ELECTROCARDIOGRAM QT CORRECTED INTERVAL PROLONGED (Investigations) | 1 (1)
ENDOCRINE DISORDERS (Endocrine disorders) | 6 (7)
EPISTAXIS (Respiratory, thoracic and mediastinal disorders) | 1 (1)
ESOPHAGITIS (Gastrointestinal disorders) | 1 (1)
EYE DISORDERS (Eye disorders) | 3 (3)
FALL (Injury, poisoning and procedural complications) | 7 (8)
FATIGUE (General disorders) | 27 (42)
FEBRILE NEUTROPENIA (Blood and lymphatic system disorders) | 1 (1)
FECAL INCONTINENCE (Gastrointestinal disorders) | 1 (1)
FEVER (General disorders) | 4 (4)
FLANK PAIN (Musculoskeletal and connective tissue disorders) | 2 (2)
FLUSHING (Vascular disorders) | 1 (1)
FRACTURE (Injury, poisoning and procedural complications) | 1 (1)
GAIT DISTURBANCE (General disorders) | 1 (1)
GASTROESOPHAGEAL REFLUX DISEASE (Gastrointestinal disorders) | 4 (4)
GASTROINTESTINAL DISORDERS (Gastrointestinal disorders) | 5 (5)
GENERAL DISORDERS AND ADMINISTRATION SITE CONDITIONS (General disorders) | 8 (17)
GENERALIZED MUSCLE WEAKNESS (Musculoskeletal and connective tissue disorders) | 1 (1)
HALLUCINATIONS (Psychiatric disorders) | 1 (1)
HEADACHE (Nervous system disorders) | 6 (6)
HEMATURIA (Renal and urinary disorders) | 11 (15)
HEMORRHOIDS (Gastrointestinal disorders) | 2 (2)
HYPERCALCEMIA (Metabolism and nutrition disorders) | 1 (1)
HYPERGLYCEMIA (Metabolism and nutrition disorders) | 19 (46)
HYPERTENSION (Vascular disorders) | 23 (44)
HYPERTHYROIDISM (Endocrine disorders) | 5 (5)
HYPERTRIGLYCERIDEMIA (Metabolism and nutrition disorders) | 1 (1)
HYPERURICEMIA (Metabolism and nutrition disorders) | 1 (1)
HYPOALBUMINEMIA (Metabolism and nutrition disorders) | 10 (15)
HYPOCALCEMIA (Metabolism and nutrition disorders) | 4 (6)
HYPOKALEMIA (Metabolism and nutrition disorders) | 14 (29)
HYPOMAGNESEMIA (Metabolism and nutrition disorders) | 19 (33)
HYPONATREMIA (Metabolism and nutrition disorders) | 5 (10)
HYPOPHOSPHATEMIA (Metabolism and nutrition disorders) | 11 (17)
HYPOTENSION (Vascular disorders) | 6 (8)
HYPOTHYROIDISM (Endocrine disorders) | 17 (20)
HYPOXIA (Respiratory, thoracic and mediastinal disorders) | 1 (1)
IMMUNE SYSTEM DISORDERS (Immune system disorders) | 1 (1)
INFECTIONS AND INFESTATIONS (Infections and infestations) | 5 (5)
INFUSION RELATED REACTION (General disorders) | 5 (7)
INFUSION SITE EXTRAVASATION (General disorders) | 1 (1)
INJURY, POISONING AND PROCEDURAL COMPLICATIONS (Injury, poisoning and procedural complications) | 1 (1)
INR INCREASED (Investigations) | 3 (3)
INSOMNIA (Psychiatric disorders) | 8 (9)
INVESTIGATIONS (Investigations) | 8 (9)
LETHARGY (Nervous system disorders) | 1 (1)
LIP INFECTION (Infections and infestations) | 1 (1)
LUNG INFECTION (Infections and infestations) | 1 (2)
LYMPHEDEMA (Vascular disorders) | 1 (1)
LYMPHOCYTE COUNT DECREASED (Investigations) | 24 (79)
MEMORY IMPAIRMENT (Nervous system disorders) | 4 (5)
METABOLISM AND NUTRITION DISORDERS (Metabolism and nutrition disorders) | 3 (3)
MUCOSITIS ORAL (Gastrointestinal disorders) | 3 (5)
MUSCLE WEAKNESS LOWER LIMB (Musculoskeletal and connective tissue disorders) | 2 (3)
MUSCULOSKELETAL AND CONNECTIVE TISSUE DISORDER (Musculoskeletal and connective tissue disorders) | 6 (9)
MYALGIA (Musculoskeletal and connective tissue disorders) | 9 (11)
MYOSITIS (Musculoskeletal and connective tissue disorders) | 1 (1)
NASAL CONGESTION (Respiratory, thoracic and mediastinal disorders) | 3 (3)
NAUSEA (Gastrointestinal disorders) | 24 (43)
NECK PAIN (Musculoskeletal and connective tissue disorders) | 3 (3)
NEOPLASMS BENIGN, MALIGNANT AND UNSPECIFIED (INCL CYSTS AND POLYPS) (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2)
NERVOUS SYSTEM DISORDERS (Nervous system disorders) | 2 (2)
NEUTROPHIL COUNT DECREASED (Investigations) | 17 (33)
NON-CARDIAC CHEST PAIN (General disorders) | 2 (2)
OBESITY (Metabolism and nutrition disorders) | 3 (4)
OSTEOPOROSIS (Musculoskeletal and connective tissue disorders) | 2 (2)
PAIN (General disorders) | 3 (3)
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 8 (9)
PALMAR-PLANTAR ERYTHRODYSESTHESIA SYNDROME (Skin and subcutaneous tissue disorders) | 2 (2)
PARESTHESIA (Nervous system disorders) | 1 (1)
PELVIC PAIN (Reproductive system and breast disorders) | 4 (5)
PERIPHERAL MOTOR NEUROPATHY (Nervous system disorders) | 1 (1)
PERIPHERAL SENSORY NEUROPATHY (Nervous system disorders) | 26 (44)
PHARYNGITIS (Infections and infestations) | 1 (1)
PLATELET COUNT DECREASED (Investigations) | 21 (58)
PLEURAL EFFUSION (Respiratory, thoracic and mediastinal disorders) | 1 (1)
PRESYNCOPE (Nervous system disorders) | 1 (1)
PRODUCTIVE COUGH (Respiratory, thoracic and mediastinal disorders) | 5 (7)
PROTEINURIA (Renal and urinary disorders) | 7 (10)
PRURITUS (Skin and subcutaneous tissue disorders) | 6 (7)
PULMONARY HYPERTENSION (Respiratory, thoracic and mediastinal disorders) | 1 (1)
RASH ACNEIFORM (Skin and subcutaneous tissue disorders) | 4 (6)
RASH MACULO-PAPULAR (Skin and subcutaneous tissue disorders) | 11 (15)
RECTAL HEMORRHAGE (Gastrointestinal disorders) | 3 (3)
RECTAL MUCOSITIS (Gastrointestinal disorders) | 1 (2)
RENAL AND URINARY DISORDERS (Renal and urinary disorders) | 7 (12)
REPRODUCTIVE SYSTEM AND BREAST DISORDERS (Reproductive system and breast disorders) | 2 (2)
RESPIRATORY, THORACIC AND MEDIASTINAL DISORDERS (Respiratory, thoracic and mediastinal disorders) | 4 (5)
RETINAL VASCULAR DISORDER (Eye disorders) | 1 (1)
SEPSIS (Infections and infestations) | 1 (1)
SINUS BRADYCARDIA (Cardiac disorders) | 1 (1)
SINUS TACHYCARDIA (Cardiac disorders) | 7 (11)
SINUSITIS (Infections and infestations) | 2 (3)
SKIN AND SUBCUTANEOUS TISSUE DISORDERS (Skin and subcutaneous tissue disorders) | 5 (7)
SKIN INFECTION (Infections and infestations) | 1 (2)
SORE THROAT (Respiratory, thoracic and mediastinal disorders) | 1 (1)
STOMACH PAIN (Gastrointestinal disorders) | 2 (2)
SYNCOPE (Nervous system disorders) | 2 (2)
THROMBOEMBOLIC EVENT (Vascular disorders) | 5 (5)
TINNITUS (Ear and labyrinth disorders) | 1 (1)
UPPER RESPIRATORY INFECTION (Infections and infestations) | 3 (3)
URINARY FREQUENCY (Renal and urinary disorders) | 3 (4)
URINARY INCONTINENCE (Renal and urinary disorders) | 3 (3)
URINARY RETENTION (Renal and urinary disorders) | 1 (1)
URINARY TRACT INFECTION (Infections and infestations) | 10 (13)
URINARY TRACT OBSTRUCTION (Renal and urinary disorders) | 1 (1)
URINARY TRACT PAIN (Renal and urinary disorders) | 6 (6)
URINARY URGENCY (Renal and urinary disorders) | 1 (3)
UTERINE HEMORRHAGE (Reproductive system and breast disorders) | 1 (1)
VAGINAL DISCHARGE (Reproductive system and breast disorders) | 1 (2)
VAGINAL DRYNESS (Reproductive system and breast disorders) | 1 (1)
VAGINAL HEMORRHAGE (Reproductive system and breast disorders) | 2 (5)
VERTIGO (Ear and labyrinth disorders) | 1 (3)
VOMITING (Gastrointestinal disorders) | 9 (11)
WATERING EYES (Eye disorders) | 2 (2)
WEIGHT GAIN (Investigations) | 1 (1)
WEIGHT LOSS (Investigations) | 14 (23)
WHEEZING (Respiratory, thoracic and mediastinal disorders) | 1 (1)
WHITE BLOOD CELL DECREASED (Investigations) | 22 (63)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol (2018-06-08): https://cdn.clinicaltrials.gov/large-docs/09/NCT02549209/Prot_000.pdf